CLINICAL TRIAL: NCT05045781
Title: Interventional, Single-ascending-dose Study Investigating the Safety, Tolerability, and Pharmacokinetic Properties of Eptinezumab in Healthy Chinese Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of Eptinezumab in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19004A
Record Dates: First submitted 2021-09-07; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Healthy
MeSH Terms: interventions — eptinezumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eptinezumab 100 mg (Experimental)
  Interventions: Drug: Eptinezumab
- Eptinezumab 300 mg (Experimental)
  Interventions: Drug: Eptinezumab

INTERVENTIONS:
Drug: Eptinezumab — single iv infusion

SUMMARY:
The purpose of the study is to investigate how the body absorbs and get rid of eptinezumab when given directly into a vein in Chinese subjects.

DETAILED DESCRIPTION:
This is an interventional, randomized, open-label, parallel-group, single-dose study investigating the safety, tolerability and pharmacokinetic properties of eptinezumab administered by intravenous (iv) infusion.

The study will consist of 20 healthy Chinese subjects, who will be randomized into two single-dose groups. The two groups will be run in parallel. In Group 1, a total of 10 subjects will receive a single iv infusion of 100 mg eptinezumab on Day 1. In Group 2, a total of 10 subjects will receive a single iv infusion of 300 mg eptinezumab on Day 1.

Safety and tolerability will be assessed throughout the study. Blood samples for plasma quantification of free eptinezumab will be collected from Day 1 to the Completion Visit (Day 84)/Withdrawal Visit.

ELIGIBILITY:
Inclusion Criteria:

* BMI of ≥ 19 and ≤ 25 kg/m2.
* The subject is Chinese, defined as being born in China and having four Chinese grandparents.
* The subject is, in the opinion of the investigator, generally healthy based on medical history, a physical examination, vital signs, an ECG, and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The subject is pregnant or breastfeeding.
* The subject has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder.

Other inclusion and exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
AUC(0-inf) eptinezumab | Day 1 to Day 84
  Area under the plasma concentration-time curve
Maximal observed plasma concentration (Cmax) of eptinezumab | Day 1 to Day 84
Systemic clearance (CL) of eptinezumab | Day 1 to Day 84
  Eptinezumab dose/AUC(0-inf)
tmax | Day 1 to Day 84
  Nominal time for the occurrence of Cmax (tmax)
Apparent terminal elimination half-life (t½) | Day 1 to Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- zs-hospital Shanghai, Shanghai, China